CLINICAL TRIAL: NCT07060911
Title: Pivotal Study to Assess Safety and Performance of Neola®, a Novel Lung Monitoring Device for Neonates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neola Medical Inc (Industry)
Responsible Party: Sponsor
Organization: Neola Medical AB (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PLN-0387
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: RDS of Prematurity; Preterm Birth; Lung Diseases
Keywords: GASMAS; Spectroscopy; Gas absorption spectroscopy
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Premature Birth; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Arm 1 (Experimental): Lung monitoring with the Neola device
  Interventions: Device: Lung monitoring with the Neola device

INTERVENTIONS:
Device: Lung monitoring with the Neola device — Lung monitoring with the Neola device

SUMMARY:
Pivotal study to assess safety and performance of Neola®, a novel lung monitoring device for neonates

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate that the device is safe and performs as intended under anticipated use conditions.

The performance of Neola will be evaluated in terms of ability to continuously measure and display the relative lung volume and absolute oxygen gas concentration during standard NICU procedures on neonates.

ELIGIBILITY:
IInclusion criteria:

* Preterm or term born neonates with gestational age between 26 and 40 weeks
* Age between 1 day post-natal and 44 weeks corrected gestational age
* Weight between 1000 g and 3500 g
* Patient treated at a neonatal intensive care unit.
* Patient is either on invasive mechanical ventilation, on CPAP or NIPPV or receives respiratory support via high-flow nasal cannula (≥2L/min)
* Signed informed consent prior to any study related procedures by the legal representatives of the patient

Exclusion criteria:

* Known cardiopulmonary congenital anomalies
* Patients with trisomies or other chromosomal abnormality
* Patients not expected to survive
* Non-intact skin or other skin conditions (such as skin lesions) that do not allow the use of skin adhesives. (e.g., Bullous impetigo, Staphylococcal scalded skin syndrome, localized lesions of herpes simplex virus)
* Thorax curvature does not allow placement of the probe sets without air between the surface of the probes and the skin.

Ages: 1 Day to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The number of device related events including skin reactions | 2 days
  The primary objective of the study is to evaluate safety with regards to adverse events (AE) and in particular device related adverse events. Outcome measure: The number of device related events including skin reactions.
The number of serious and non-serious adverse events occurring during the trial | 2 days
  The primary objective of the study is to evaluate safety with regards to adverse events (AE) and in particular device related adverse events. Outcome measure: The number of serious and non-serious adverse events occurring during the trial.

SECONDARY OUTCOMES:
The device's ability to continuously measure and present the clinical parameters while the neonates are in a resting state/sleeping | 7 days
  This endpoint will be presented as the percentage of the total resting/sleeping time that the device is able to measure the clinical parameters relative lung volume and absolute oxygen concentration.
The device's ability to continuously measure and present the clinical parameters during normal handling of the neonates | 7 days
  This endpoint will be presented as the percentage of the total handling time that the device is able to measure the clinical parameters relative lung volume and absolute oxygen concentration.
The adhesive performance of the probes in terms of ability to be repositioned and stay attached | 7 days
  The adhesive performance of the probes in terms of ability to be repositioned and stay attached. This exploratory endpoint will be evaluated the percentage of probe adhesives that were able to stay attached for the duration of the measurement session

OTHER OUTCOMES:
Evaluate the correlation between Neola® measured clinical data and clinical data available from other monitoring devices, procedures or tests. | 7 days
  The endpoint will be valuated using diagnostic methods such as, but not limited to: peripheral oxygen saturation (SpO2), x-ray images, Blood gas analysis data (partial pressure of oxygen (PaO2) and carbon dioxide (PaCO2)), respiratory support settings, respiratory rate, heart rate, blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Chock, M.D., M.S. Epi, Principal Investigator — Division of Neonatal and Developmental Medicine Stanford University School of Medicine; Vineet Bhandari, MD, DM, Principal Investigator — Department of Pediatrics The Children's Regional Hospital at Cooper
Locations (2):
- United States (2):
  - Stanford Lucile Packard Children's Hospital Neonatal Intensive Care Unit, Palo Alto, California
  - Cooper Health System, Camden, New Jersey

IPD SHARING:
Plan to Share IPD: No